CLINICAL TRIAL: NCT05667012
Title: Effect of an Online Education Program Through Information Pills in Women Who Practice Sports for the Prevention of Stress Urinary Incontinence
Brief Title: Online Education Program in Sportswomen for the Prevention of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ED_IU_ONLINE
Record Dates: First submitted 2022-12-14; First posted 2022-12-28 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Incontinence Stress
Keywords: Educational pills; Prevention; Sports; Physiotherapy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator analyzing the results will be blinded to the intervention group to which the participants belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity (Experimental): Women who practice sports professionally.
  Interventions: Other: Educational videos
- Low intensity (Active Comparator): Women who practice sport in a non-professional way.
  Interventions: Other: Educational videos

INTERVENTIONS:
Other: Educational videos — There will be a total of 6 videos, each of these videos will last between 8 and 10 minutes and will be accessed through a YouTube link to a private channel.

SUMMARY:
Stress urinary incontinence (SUI) can be defined through its symptoms as the involuntary loss of urine when carrying out an activity or effort that implies an increase in intra-abdominal pressure (IAP).

Perineal dysfunctions are a widespread problem among the sportswomen population. Therefore, a continuous exposure to exercises that entail a high intra-abdominal pressure such as that which occurs in high-impact sports in women.

As seen in other studies in which pelvic floor educational programs were taught; advice and guidance focused on perineal health education helped participants improve knowledge, symptoms, and quality of life, as well as reduce the incidence of SUI.

For these reasons, it is relevant to carry out a prevention and education program in the female population who play high-impact sports, since they have a high prevalence of SUI.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) can be defined through its symptoms as the involuntary loss of urine when carrying out an activity or effort that implies an increase in intra-abdominal pressure (IAP), for example, coughing, sneezing or performing sports activities that involve hyperpressive gestures.

Perineal dysfunctions are a widespread problem among the population. Within these dysfunctions, the presence of stress urinary incontinence can be highlighted, the incidence of which is higher in women. Among its risk factors the investigators find; advanced age, obesity, gynecological surgery, pregnancy and vaginal delivery (increasing the risk if it is an instrumental delivery).

On the other hand, although the practice of regular exercise and having an active life is a protective factor for a good physical-functional state, a continuous exposure to exercises that entail a high intra-abdominal pressure such as that which occurs in high-impact sports in women, is another important risk factor to take into account in this population. Of the risk factors, the practice of high-impact sports has also been found, so one in four women who practice different sports classified as high-impact have also ended up developing this pathology.

In addition to the problems at the functional level that SUI entails, the impact it has on the quality of life of the people who suffer from it should be emphasized, assuming the patients feelings related to low mood, frustration, discomfort, modesty, etc. Therefore, their work, social and personal lifestyle is also altered.

In other studies in which pelvic floor educational programs were taught; advice and guidance focused on perineal health education helped participants improve knowledge, symptoms, and quality of life, as well as reduce the incidence of SUI. This is where physiotherapists intervene, since they have an essential role in the transmission of information regarding its prevention and treatment.

For these reasons, it is relevant to carry out a prevention and education program in the female population who play high-impact sports, since they have a high prevalence of SUI, as recommended by the seventh professional principle applied to physiotherapy. Education about the perineal sphere in women reduces the practice of habits that may put their pelvic floor at risk. Despite this, currently in primary care there are not a large number of programs for perineal health. This is demonstrated by different investigations that maintain that almost all the women who participated in them had not consulted their symptoms with anyone or had heard of the pelvic floor muscles or strengthening exercises. Without forgetting that it is increasingly common for women to be present in sports at a professional level, where their demands can favor the increase in the prevalence of suffering from SUI. For this reason, this study intends to observe the effects of a SUI prevention program in female athletes, both low and high level, and check whether there are differences at both levels.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 35 years old.
* For the control group who have done sports at least 2 days a week for at least 1 year.
* For the experimental group who are semi or professional athletes and who carry out high intensity/impact.

Exclusion Criteria:

* Pregnant or postpartum women or who have undergone gynecological and/or urogynecological surgeries.
* Respiratory, musculoskeletal, metabolic and neurological diseases.
* A minimum of MMS>21.
* Refusal to participate or incomplete questionnaires.
* That they have not been diagnosed with UI of any cause.
* No mastery or comprehension of the Spanish language.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge | 0 week (baseline)
  The validated Spanish PIKQ questionnaire will be used. This questionnaire has good validity and reliability. It is structured in 13 questions with closed answers, that is, "I agree" or "I disagree" answers. These questionnaires evaluate items about UI and prolapses, mainly. Your scoring range is 0 to 1. On each scale, the minimum score is 0 and the maximum is 12.
Knowledge | 4 week
  The validated Spanish PIKQ questionnaire will be used. This questionnaire has good validity and reliability. It is structured in 13 questions with closed answers, that is, "I agree" or "I disagree" answers. These questionnaires evaluate items about UI and prolapses, mainly. Your scoring range is 0 to 1. On each scale, the minimum score is 0 and the maximum is 12.

SECONDARY OUTCOMES:
Motivation | 0 week (pre), 4 week (post)
  For the perception of exercise, the Markland and Tobin (2004) behavior regulation scale for physical exercise (BREQ-2) will be used. It consists of 19 items, which are answered according to a 5-point Likert-type scale ranging from 0 to (strongly disagree) to 4 (strongly agree), grouped into five factors: demotivation (4 items: e.g., "I don't see the point of exercising"), external regulation (4 items: e.g., "I exercise to pleasing other people"), introjected regulation (3 items: e.g., "I exercise because I feel guilty when I don't practice"), identified regulation (3 items: e.g., "I exercise because I value the benefits of physical exercise ") and intrinsic regulation (4 Items: e.g., "I exercise because I think exercise is fun").
Perception | 0 week (pre), 4 week (post)
  The perception of change after the intervention was measured using the Patient Global Impression of Change (PGIC) validated in Spanish. This test reflects the patient's belief about the effect of the applied treatment. A scale is used that goes from 1 (the patient is much better) to 7 (the patient is much worse). It also consists of a visual analogue scale that ranked the improvement from 0 to 10, with the first value being a very good improvement and the second being a significant worsening after treatment.
Quality of life of participants | 0 week (pre), 4 week (post)
  To test the quality of life, the validated questionnaire in Spanish EQ-5D will be used. This is made up of 5 questions with five options and an analog scale from 1 to 100. In this, both physical capacities, such as pain, anxiety and health level.
Adherence | 0 week (pre), 4 week (post)
  To know the adherence of the patients, a record will be kept of the number of views of each video by group.
Sexual function | 0 week (pre), 4 week (post)
  To test female sexual function we use the FSFI Questionnaire. This contains 19 questions about sexuality during the last 4 weeks, referring to sexual desire or interest, sexual arousal and satisfaction, among other things. The subscales have a range from 0 (or 1) to 5 (higher scores indicate better sexual function).
Satisfaction after the intervention | 0 week (pre), 4 week (post)
  A questionnaire of 4-5 questions will be passed in order to collect the satisfaction of the participants after the intervention. Each question will have 5 multiple choices ranging from "strongly disagree" to "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández Guillén, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy of the University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuentes-Aparicio L, Dominguez-Navarro F, Maudos-Soriano A, Hernandez-Guillen D. eHealth educational intervention: effects of an online video program in prevention of the pelvic women's health-a non-randomized experimental study. Arch Gynecol Obstet. 2025 Dec;312(6):2153-2164. doi: 10.1007/s00404-025-08200-6. Epub 2025 Oct 3. PMID 41042325